CLINICAL TRIAL: NCT01035944
Title: Evaluation of Use of Chitosan-Based Dressings to Facilitate Safe, Effective Debridement of Chronic Wounds in Operating Room and Inpatient Ward and Minimize Bacterial Re-Colonization of Wounds.
Brief Title: Chitosan Dressings to Facilitate Safe Effective Debridement of Chronic Wounds & Minimize Wound Bacterial Re-colonization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet enrollment milestones
Sponsor: HemCon Medical Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC-NU-2009-01
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-05

CONDITIONS: Wound Debridement
Keywords: Chronic wounds; Chronic wound debridement; Debridement; Bedside debridement; Surgical debridement; Wound debridement; Minimize bacterial re-colonization of wounds; HemCon ChitoGauze Dressings; HemCon Dressings; Chitosan-based dressings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HemCon Operating Room (Experimental): The HemCon dressing is the intervention for the HemCon Operating Room arm. The first sub-study will evaluate the use of HemCon dressings in the operating room setting. 20 patients will be treated with HemCon dressings following a debridement, and 20 patients will be treated with gauze dressings following a debridement.
  Interventions: Device: HemCon Dressings and HemCon ChitoGauze; chitosan-based.
- Control Operating Room (Active Comparator): The first sub-study will evaluate the use of HemCon dressings in the operating room setting. 20 patients will be treated with HemCon dressings following a debridement, and 20 patients will be treated with gauze dressings following a debridement.
  Interventions: Device: Gauze and saline dressings.
- HemCon Bedside (Experimental): The intervention for the HemCon Beside arm is the HemCon Dressing. The other sub-study will evaluate the use of HemCon dressings compared to control dressings in bedside debridement. In this sub-study, 20 patients will be treated with HemCon dressings following a debridement, and 20 patients will be treated with gauze dressings following a debridement.
  Interventions: Device: HemCon Dressings and HemCon ChitoGauze; chitosan-based.
- Control Bedside. (Active Comparator): The other sub-study will evaluate the use of HemCon dressings compared to control dressings in bedside debridement. In this sub-study, 20 patients will be treated with HemCon dressings following a debridement, and 20 patients will be treated with gauze dressings following a debridement.
  Interventions: Device: Gauze and saline dressings.

INTERVENTIONS:
Device: HemCon Dressings and HemCon ChitoGauze; chitosan-based. — Perform debridement of chronic wounds using HemCon chitosan-based dressings and HemCon ChitoGauze both at bedside and in the Operating Room (OR) settings. Control for both settings will be gauze and saline dressings.
  Other Names: HemCon Dressings, HemCon ChitoGauze.
  Arms: HemCon Bedside; HemCon Operating Room
Device: Gauze and saline dressings. — Control for both settings will be gauze and saline dressings.
  Arms: Control Bedside.; Control Operating Room

SUMMARY:
The purpose of this study is to determine if the use of HemCon chitosan-based dressings is effective to facilitate safe, effective debridement of chronic wounds in the operating room and inpatient ward settings and to minimize bacterial re-colonization of wounds.

DETAILED DESCRIPTION:
Primary objective: There are two primary objectives:

1. To demonstrate that debridements performed using HemCon dressings at the bedside can be performed safely without excessive bleeding in eligible patients
2. To compare the levels of bacterial load between debrided wounds treated with HemCon dressings and debrided wounds treated with gauze and saline dressings at 2 days and 5 days after debridement

Secondary objectives: The following secondary objectives will be achieved by this study:

1. To determine the cost efficacy, if any, between wounds debrided at the bedside with HemCon dressings and wounds debrided in the operating room setting
2. To determine the cost efficacy, if any, between wounds debrided in the operating room where hemostasis is achieved with a HemCon dressing and between debrided wounds where hemostasis is achieved with traditional cauterization methods.
3. To compare comfort levels in patients treated with HemCon dressings as compared to traditional gauze dressings.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and are able to provide written informed consent.
* Have a wound on their body with an eschar and/or significant slough present
* Documented laboratory studies and coagulation profiles prior to the debridement (including hematocrit, hemoglobin, white blood count, total lymphocyte count, albumin, pre-albumin, HbA1C in patients with diabetes)
* Subjects with a hemoglobin < 9 g/dL must have one unit of blood typed and cross matched prior to the debridement; all other subjects must have an active type and screen performed prior to the debridement procedure.
* Subjects must be willing to consent to a blood transfusion in the rare event that a transfusion is necessary.
* Must be expected to be inpatients for at least 5 days following debridement, to enable controlled dressing changes by the service.
* Female subjects of childbearing age must not be pregnant, and must consent to utilize an appropriate method of contraception during the course of the study.

For subjects that are to undergo a debridement in the operating room:

* Subjects must be sensate or have wounds that are sufficiently large to warrant a debridement in the OR
* Wounds must require more than a simple eschar removal, or must be extensive enough that an operating room debridement would be more appropriate.
* Subjects must be candidates for regional or general anesthesia, unless the wound occurs in an insensate body part (for example, a pressure sore in a paraplegic or quadriplegic patient, or a diabetic foot ulcer in a patient with a dense diabetic polyneuropathy).

For subjects that are to undergo a debridement in the bedside setting:

* The part of the wound that is to be debrided must be mostly an eschar and necrotic tissue which is not likely to have significant bleeding.
* Subjects must be insensate, or the wound must be less than 50 cm2 such that the use of local anesthesia in the wound can be undertaken.

Exclusion Criteria:

* Pre-debridement hemoglobin level < 7.0 g/dL
* Not candidates for or refuse blood transfusions
* Unable to provide written informed consent
* Subjects with sensitivity to chitosan or the gauze dressings used in this study, or any local anesthetic needed for a debridement
* Subjects who are in the intensive care unit
* Subjects who, in the opinion of the Investigator, may not complete the study for any reason.
* Have grossly infected wounds that may reasonably be expected to require multiple debridement procedures prior to clearance of bacteria and nonviable tissue from the wound.
* For wounds situated in the lower extremity, leg must have either palpable pulses or else an ABI > 0.4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Galiano, M.D., Principal Investigator — Northwestern Memorial Hospital, Division of Plastic Surgery
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HemCon Operating Room | Control Operating Room | HemCon Bedside | Control Bedside.
Started | 14 | 14 | 5 | 4
Completed | 11 | 13 | 4 | 4
Not Completed | 3 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HemCon Operating Room | Control Operating Room | HemCon Bedside | Control Bedside. | Total
Number analyzed (Participants) | 14 | 14 | 5 | 4 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.43 (20.0) | 51.64 (16.2) | 70.80 (19.9) | 64.50 (20.8) | 57.05 (19.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 2 | 3 | 22
  Male | 4 | 7 | 3 | 1 | 15
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 5 | 4 | 37

OUTCOME MEASURES:

1. Primary Outcome: Demonstrate That Debridements Using HemCon Dressings at Bedside Can be Performed Safely Without Excessive Bleeding; Compare Levels of Bacterial Load Between Debrided Wounds Treated With HemCon Dressings vs. Wounds Treated With Gauze & Saline Dressings.
Time Frame: 2 days and 5 days after debridement.
Population: Zero participant data were analyzed. Study was terminated early; unable to reach enrollment milestones.
Arm/Group | HemCon Operating Room | Control Operating Room | HemCon Bedside | Control Bedside.
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Determine Cost Efficacy, Hemostasis and Patient Comfort Between Wounds Debrided at Bedside With HemCon Dressings & Wounds Debrided in Operating Room Setting.
Time Frame: 2 days and 5 days after debridement.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | HemCon Operating Room | Control Operating Room | HemCon Bedside | Control Bedside.
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 2/14 | 1/14 | 1/5 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HemCon Operating Room (N=14) | Control Operating Room (N=14) | HemCon Bedside (N=5) | Control Bedside. (N=4)
Acute Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Stroke (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bleeding Wound (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Significant amount of bacteria in wound (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
transfusion reaction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound hematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the study; unable to reach enrollment milestones. No outcome measure data was analyzed; zero participants were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less